CLINICAL TRIAL: NCT04586985
Title: A Phase 1 Randomized, Double-Blind, Placebo-Controlled, Single-and Multiple-Dose Study Evaluating Safety, Tolerability, and Pharmacokinetics, With an Open-Label Initial Food Effect and CYP3A Drug-Drug Interaction Study, of FTX-6058 in Healthy Adult Subjects, and a Randomized, Double-Blind, Placebo-Controlled Multiple-Dose Study Evaluating, Safety, Tolerability and Pharmacokinetics in Subjects With Sickle Cell Disease (SCD)
Brief Title: Safety, Tolerability and Pharmacokinetics of FTX-6058
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Fulcrum Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FIS-002-2020
Record Dates: First submitted 2020-10-05; First posted 2020-10-14 (Actual); Last update posted 2022-12-12 (Actual); Status verified 2022-12

CONDITIONS: Healthy Adult Subjects; Sickle Cell Disease
Keywords: Healthy Adult Subjects; Sickle Cell Disease; Sickle Cell Anemia; Sickle Cell Disorder
MeSH Terms: conditions — Anemia, Sickle Cell

STUDY DESIGN:
Intervention Model Description: Single ascending dose escalation and multiple ascending dose escalation study followed by an evaluation of food effects on absorption and CYP3A induction
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Randomized double-blind, placebo-controlled
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Single Ascending Dose (SAD) cohorts in Healthy Subjects (Part A) (Experimental): Subjects will be randomized to receive a single dose of FTX-6058 or placebo. Cohorts 1 and 2 will enroll 5 subjects per cohort randomized 3:2. Cohorts 3-8 will enroll 7 subjects per cohort randomized 5:2. Planned doses are 2 mg (Cohort 1), 4 mg (Cohort 2), 10 mg (Cohort 3), 20 mg (Cohort 4), 30 mg (Cohort 5), 40 mg (Cohort 6), 60 mg (Cohort 7), and 90 mg (Cohort 8).
  Interventions: Drug: FTX-6058/placebo oral capsule(s)
- Multiple Ascending Dose (MAD) cohorts in Healthy Subjects (Part B) (Experimental): Subjects will be randomized 3:1 to receive once daily FTX-6058 or placebo by mouth for 14 days. Up to 6 cohorts of 8 subjects per cohort will be enrolled. Planned doses are 2 mg (Cohort 1), 6 mg (Cohort 2), 10 mg (Cohort 3), 20 mg (Cohort 4), 30 mg (Cohort 5), and 40 mg (Cohort 6).
  Interventions: Drug: FTX-6058/placebo oral capsule(s)
- Pilot Food Effect Cohort in Healthy Subjects (Part C) (Experimental): Ten subjects will be randomized to receive a single 20 mg dose of FTX-6058 with and without a high-fat meal with a washout period of 4 days.
  Interventions: Drug: FTX-6058 - Two Dosing Periods
- Potential for CYP3A Induction in Healthy Subjects (Part D) (Experimental): Sixteen subjects will receive 3 mg Midazolam once by mouth on Day 1. On Days 3-12, subjects will receive FTX-6058 by mouth once daily. On Day 12, a second dose of 3 mg Midazolam will be given once by mouth. The dose of FTX-6058 will be the highest tolerated dose from Part B.
  Interventions: Drug: FTX-6058 / Midazolam Syrup
- Multiple Dose Cohort in Sickle Cell Disease Subjects (Part E) (Experimental): Subjects will be randomized 3:1 to receive FTX-6058 or placebo once daily by mouth for 14 days. Up to 8 subjects will be enrolled. The planned dose is 6mg.
  Interventions: Drug: FTX-6058/placebo oral capsule(s)

INTERVENTIONS:
Drug: FTX-6058/placebo oral capsule(s) — Subjects will receive FTX-6058 or matching placebo.
  Arms: Single Ascending Dose (SAD) cohorts in Healthy Subjects (Part A)
Drug: FTX-6058/placebo oral capsule(s) — Subjects will receive FTX-6058 or matching placebo.
  Arms: Multiple Ascending Dose (MAD) cohorts in Healthy Subjects (Part B)
Drug: FTX-6058 - Two Dosing Periods — Subjects will receive FTX-6058
  Arms: Pilot Food Effect Cohort in Healthy Subjects (Part C)
Drug: FTX-6058 / Midazolam Syrup — Subjects will receive FTX-6058 and midazolam syrup
  Arms: Potential for CYP3A Induction in Healthy Subjects (Part D)
Drug: FTX-6058/placebo oral capsule(s) — Subjects will receive FTX-6058 or matching placebo.
  Arms: Multiple Dose Cohort in Sickle Cell Disease Subjects (Part E)

SUMMARY:
This is a study to evaluate the safety, tolerability and pharmacokinetics of FTX-6058 in healthy adult subjects and adult subjects with sickle cell disease (SCD).

DETAILED DESCRIPTION:
This study is a Phase 1 randomized, double-blind, placebo-controlled, single- and multiple-dose study evaluating safety, tolerability, and pharmacokinetics, with an open-label initial food effect and CYP3A drug-drug interaction study, of FTX-6058 in healthy adult subjects and a randomized, double-blind, placebo-controlled, multiple-dose study in adult subjects with sickle cell disease (SCD).

This study will comprise 5 parts and will be conducted in healthy adult subjects and adult subjects with sickle cell disease (SCD) (Part E only).

Part A will be a randomized, double-blind, placebo-controlled, single ascending dose (SAD) study in up to 8 cohorts of healthy adult subjects. Part B will be a randomized, double-blind, placebo-controlled, multiple ascending dose (MAD) study in up to 6 cohorts of healthy adult subjects dosed once daily for 14 days. Part C will be an open-label pilot food effect study in healthy adult subjects randomized to take FTX-6058 with and without a high-fat meal, and Part D will be an open-label study to evaluate the potential of FTX-6058 to induce CYP3A (using midazolam) in healthy adult subjects. Part E will be a randomized, double-blind, placebo-controlled, multiple dose study in adult subjects with sickle cell disease (SCD). Subjects in Part E may enroll into Study 6058-SCD-101 (NCT 05169580) Part A (6 mg cohort) at the Day 15 visit; subjects that enroll into 6058-SCD-101 will not need to undergo the Safety Follow-up visit.

The primary endpoint of the study is to evaluate the safety and tolerability of FTX-6058 in healthy adult subjects and adult subjects with sickle cell disease as measured by the frequency of adverse events. Secondary endpoints include evaluation of the pharmacokinetics of single dose and multiple dose FTX-6058 in healthy adult subjects, pharmacokinetics of multiple dose FTX-6058 in adult subjects with sickle cell disease, evaluation of the potential effect of food on FTX-6058 and evaluation of the potential for CYP3A induction by FTX-6058 in healthy adult subjects.

ELIGIBILITY:
Inclusion Criteria: Healthy Subjects

1. Healthy male / female subjects, 18 to 55 years of age, inclusive at screening.
2. Good health, based upon the opinion of the investigator and the results of medical history, physical examination, vital signs, ECG, and laboratory profiles of both blood and urine at screening.
3. Body mass index (BMI) between 18 and 32 kg/m², inclusive at screening, and with a minimum weight of 50 kg.
4. Willingness of men and women of reproductive potential to agree to use two effective means of contraception throughout study participation until 90 days after dose administration.
5. Signed and dated written informed consent.
6. Willing and able to comply with all study procedures.
7. Females with hematocrit >35% and <45% or hemoglobin >11.7/dL and <15.5/dL and males with hematocrit >38.5% and <50% or hemoglobin >13.2/dL and <17.1/dL.

Exclusion Criteria: Healthy Subjects

1. History of any illness or any clinical condition that, in the opinion of the investigator/sub-investigator, might confound the results of the study or pose an additional risk in administering study drug to the subject. This may include, but is not limited to, history or presence of gastrointestinal conditions including Crohn's disease, ulcerative colitis, frequent episodes of diarrhea, or irritable bowel syndrome; history of relevant drug or food allergies; history of cardiovascular or central nervous system disease; history or presence of clinically significant pathology; clinically significant history of mental disease; concurrent active malignancy; and history of cancer, except for squamous cell skin cancer, basal cell skin cancer, and Stage 0 cervical carcinoma in situ (all 3 with no recurrence for the last 5 years).
2. History of febrile illness within 1 week prior to the baseline visit.
3. Acute or chronic history of liver disease or current alanine aminotransferase ≥ 2 × ULN or total bilirubin >1.5 × ULN at screening (Note: Subjects with Gilbert's syndrome are permitted to enroll in the trial).
4. Known renal impairment (defined as glomerular filtration rate of <60 mL/min/1.73 m²).
5. Positive screen for hepatitis B surface antigen (HBsAg), hepatitis C virus (HCV) antibody, or antibodies against human immunodeficiency viruses 1 and 2 (HIV1/HIV2 Abs) at screening.
6. Any condition possibly affecting drug absorption (e.g., gastrectomy, cholecystectomy, or other gastrointestinal tract surgery, except appendectomy).
7. Standard 12 lead ECG demonstrating QTcF >450 msec for male subjects and QTcF >470 msec for female subjects at screening. If QTcF exceeds 450 msec for males or 470 msec for females, the ECG will be repeated 2 more times, and the average of the 3 QTcF values will be used to determine the subject's eligibility.
8. History of cardiac dysrhythmias requiring anti-arrhythmia treatment(s) or history or evidence of abnormal ECGs that, in the opinion of the investigator or medical monitor, would preclude the subject's participation in the study.
9. Blood or blood product (e.g., plasma/serum) donation (of approximately 1 pint [500 mL] or more) or any significant loss of blood within 8 weeks prior to screening or intention to donate blood or blood products during the study as determined by the investigator.
10. History of abuse of addictive substances such as drug abuse, or regular user of sedatives, hypnotics, tranquilizers, or any other addictive agent within 6 months prior to screening.
11. History of regular alcohol consumption within 6 months prior to screening defined as: (a) An average weekly intake of greater than 21 units. One unit is equivalent to a 285 mL glass of full-strength beer or 425 mL of light beer or 1 (30 mL) measure of spirits or 1 glass (100 mL) of wine.
12. History of demonstrating an excess in xanthine or caffeine consumption (more than 8 cups of coffee or equivalent per day).
13. Use of another investigational product within 30 days or 5 half-lives (whichever is longer), or according to local regulations, or currently participating in a prospective study with an investigational product or medical device.
14. Use of any medication (prescription or over-the-counter [OTC]) within 14 days of study drug administration, or use of herbal supplements, dietary supplements or multivitamins within 7 days of study drug administration or less than 5 half-lives (whichever is longer), with the exception of paracetamol (up to 3 g/day). Other exceptions will only be made if the rationale is clearly documented by the investigator (a) Note: Any vaccination, including COVID-19 vaccine, cannot be administered within 14 days prior to initial dose of study drug until the end of study participation.
15. History of sensitivity to the study drug or placebo, or a history of drug or other allergy that, in the opinion of the investigator or medical monitor, contraindicates their participation.
16. Female subject who is pregnant, trying to become pregnant, or is breastfeeding or male subject whose partner is pregnant, trying to become pregnant, or is breastfeeding.
17. Subject is mentally or legally incapacitated.
18. Abnormal laboratory results indicative of any significant medical disease that, in the opinion of the investigator, would preclude the subject's participation in the study at screening or prior to first dose.
19. Subject, or close relative of the subject, is the investigator or a sub-investigator, research assistant, pharmacist, study coordinator, or other staff directly involved with the conduct of the study at that site.
20. Positive test for drugs of abuse at screening or baseline.
21. Positive test for COVID-19 prior to admission to the study site, as required per local regulations.
22. Subject smokes cigarettes (or equivalent) and/or has used nicotine-based products within 3 months prior to screening. (a) Note: Cotinine test is not required per protocol but may be performed at the discretion of the Investigator to confirm non-smoker status.
23. Consumption of any alcohol within the 48-hour period prior to study drug administration.
24. Plans for hospitalization, surgery, or other major procedures during the study duration or between screening and baseline.
25. Part D Only: Any contraindication to the use of midazolam.

Inclusion Criteria: Sickle Cell Disease Subjects

1. Subject is 18 to 55 years of age at the time informed consent is obtained. Subject has provided consent before any study-specific procedures are performed and is willing and able to comply with the study procedures and restrictions.
2. Body mass index (BMI) between 18 and 32 kg/m², inclusive at screening, and with a minimum weight of 50 kg
3. Willingness of men and women of reproductive potential must agree to use 2 effective means of contraception throughout study participation until 90 days after dose administration.
4. Signed and dated written informed consent.
5. Confirmed Sickle Cell Disease (SCD) at the time of screening (SS and S/β⁰) by high performance liquid chromatography (HPLC).
6. HbF ≤20% of total hemoglobin (Hb) at screening by HPLC
7. SCD characterized by both of the following: (a) Total hemoglobin between 5.5 and 10.5 g/dL at screening; (b) 0-6 vaso-occlusive crisis (VOC) episodes over the 12 months prior to screening (VOC is defined as pain crises (defined as an acute onset of pain for which there is no other medically determined explanation other than vaso- occlusion and which requires therapy with oral or parenteral opioids or parenteral NSAIDs) as well as other complicated crises, such as acute chest syndrome (ACS), priapism, and hepatic or splenic sequestration.).
8. Subject must meet both of the following laboratory values at screening: (a) Absolute neutrophil count ≥1.5/ × 10⁹/L; (b) Platelets ≥80 × 10⁹/L
9. Absolute reticulocyte count at screening higher than 100 × 10⁹/L

Exclusion Criteria: Sickle Cell Disease Subjects

1. Major surgery, hospitalization, infection, significant bleeding, cerebrovascular accident or seizure, or transfusion within 14 days prior to study enrollment through conclusion of study follow-up period; elective surgery planned for the time period of the trial.
2. Sickle cell complication requiring hospitalization in the past 14 days or > 6 total VOCs over the past 12 months requiring hospitalization.
3. Use of opioids and/or opiates (unless used for chronic pain management), anticoagulants, or medications that induce or inhibit CYP3A4 within 14 days prior to starting study drug or anticipated need for any of these agents during the study. (Pain meds for chronic pain management or VOC events occurring during the study may be administered at the discretion of the investigator.)
4. Use of voxelotor or hydroxyurea within 60 days prior to starting study drug.
5. Participation in any other investigative treatment studies within the past 60 days.
6. History of bone marrow transplant or human stem cell transplant or gene therapies.
7. Vaccination (including against COVID-19) in the previous 14 days.
8. Positive test for COVID-19 prior to admission to the study site, as required per local regulations.
9. Significant abnormalities in hepatic biochemical tests that, in the opinion of the investigator, are outside the typical range seen with SCD. Potential subjects are to be excluded if alanine aminotransferase (ALT) or aspartate transaminase (AST) ≥3× ULN or albumin <2.0 mg/dL or direct (conjugated) bilirubin ≥1.5 mg/dL or prothrombin time/international normalized ratio > 1.5 ULN.
10. Subjects with end stage renal disease defined as glomerular filtration rate <10 mL/min/1.73m², using Schwartz formula or serum creatinine >1.2 mg/dL and calculated creatinine clearance <30 mL/min. Subjects on dialysis are excluded.
11. Subjects with abnormal laboratory results indicative of any significant medical disease that, in the opinion of the investigator, would preclude the subject's participation in the study or potentially obscure the interpretation of the scheduled assessments. Screening laboratory assessments may be repeated up to twice at the discretion of the investigator.
12. Subjects being treated with antiretroviral agents (such as didanosine and stavudine).
13. Infection with human immunodeficiency virus (HIV), hepatitis B, or hepatitis C such that subjects are currently on therapy or will be placed on therapy during the trial
14. Subjects receiving regularly scheduled transfusions to reduce levels of HbS.
15. Clinically diagnosed substance use disorder for alcohol or other illicit drugs of abuse. Positive urine drug screen at screening or on day of admission for substances other than marijuana or prescribed opioids/opiates for chronic pain management is exclusionary.
16. Pregnant or lactating female; or female of childbearing age unable or unwilling to comply with birth control or abstinence during the course of the study.
17. Febrile illness in the 7 days prior to baseline visit.
18. Subject is investigative site personnel or member of their immediate family (spouse, parent, child or sibling whether biological or legally adopted).
19. Heart rate corrected QT interval-Frederica's method (QTcF) >450 msec male and >470 msec female.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 109 (Actual)
Dates: Start 2020-10-26 (Actual); Primary Completion 2022-11-15 (Actual); Study Completion 2022-11-15 (Actual)

PRIMARY OUTCOMES:
Treatment-Emergent Adverse Events | Up to approximately 4 weeks of monitoring
  To evaluate the safety and tolerability of FTX-6058 in healthy adult subjects and adult subjects with sickle cell disease based on the frequency of adverse events (AEs), frequency of serious adverse events (SAEs), and clinically significant laboratory test results, electrocardiograms (ECGs), and vital signs.

SECONDARY OUTCOMES:
Plasma Concentrations of FTX-6058 | Study Part A: Days 1, 2, 3 and 4
  Blood samples will be collected to measure the plasma concentration of FTX-6058 at specified timepoints by liquid chromatography with tandem mass spectrometry.
Plasma Concentrations of FTX-6058 | Study Part B: Days 1, 2, 7, 8-10, 11-14 and 15
  Blood samples will be collected to measure the plasma concentration of FTX-6058 at specified timepoints by liquid chromatography with tandem mass spectrometry
Plasma Concentrations of FTX-6058 | Study Part C: Days 1-4
  Blood samples will be collected to measure the plasma concentration of FTX-6058 at specified timepoints by liquid chromatography with tandem mass spectrometry.
Plasma Concentrations of Midazolam | Study Part D: Days 1, 2, 12 and 13
  Blood samples will be collected to measure the plasma concentration of Midazolam at specified timepoints by liquid chromatography with tandem mass spectrometry
Plasma Concentrations of for 1-OH-Midazolam | Study Part D: Days 1, 2, 12 and 13
  Blood samples will be collected to measure the plasma concentration of 1-OH-Midazolam at specified timepoints by liquid chromatography with tandem mass spectrometry.
Plasma Concentrations of FTX-6058 | Study Part E: Days 1, 7 and 14
  Blood samples will be collected to measure the plasma concentration of FTX-6058 at specified timepoints by liquid chromatography with tandem mass spectrometry.

OTHER OUTCOMES:
Predictive Model of the Relationship between FTX-6058 Concentration and QTc Intervals | Study Part A: Days 1 and 2
  A model of the relationship between time-match FTX-6058 plasma concentrations and QTc intervals may be developed and will include simulations to predict potential QT risk.
Predictive Model of the Relationship between FTX-6058 Concentration and QTc Intervals | Study Part B: Days 1, 2, and 7-15
  A model of the relationship between time-match FTX-6058 plasma concentrations and QTc intervals may be developed and will include simulations to predict potential QT risk.
Target Engagement of FTX-6058 | Study Part B: Days -1, 7, 11-14 and 7-10 days after last dose of study drug
  Change from baseline in H3K27me3/Total Histone H3 ratio in circulating monocytes will be evaluated by fluorescence-activated cell sorting (FACS).
Target Engagement of FTX-6058 | Study Part E : Days -1, 7,14 and and 7-10 days after last dose of study drug
  Change from baseline in H3K27me3/Total Histone H3 ratio in circulating monocytes will be evaluated by fluorescence- activated cell sorting (FACS).

CONTACTS AND LOCATIONS:
Overall Officials: John Ziegler, MD, FASA, Study Director — Fulcrum Therapeutics
Locations (2):
- United States (2):
  - Atlanta Center for Medical Research - Sickle Cell Subjects Only, Atlanta, Georgia
  - Altasciences Clinical Kansas, Inc. - Healthy Adults Subjects Only, Overland Park, Kansas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ngo DA, Aygun B, Akinsheye I, Hankins JS, Bhan I, Luo HY, Steinberg MH, Chui DH. Fetal haemoglobin levels and haematological characteristics of compound heterozygotes for haemoglobin S and deletional hereditary persistence of fetal haemoglobin. Br J Haematol. 2012 Jan;156(2):259-64. doi: 10.1111/j.1365-2141.2011.08916.x. Epub 2011 Oct 24. PMID 22017641
- [Background] Piel FB, Steinberg MH, Rees DC. Sickle Cell Disease. N Engl J Med. 2017 Apr 20;376(16):1561-1573. doi: 10.1056/NEJMra1510865. No abstract available. PMID 28423290
- [Background] Sankaran VG, Orkin SH. The switch from fetal to adult hemoglobin. Cold Spring Harb Perspect Med. 2013 Jan 1;3(1):a011643. doi: 10.1101/cshperspect.a011643. PMID 23209159
- [Background] Saraf SL, Molokie RE, Nouraie M, Sable CA, Luchtman-Jones L, Ensing GJ, Campbell AD, Rana SR, Niu XM, Machado RF, Gladwin MT, Gordeuk VR. Differences in the clinical and genotypic presentation of sickle cell disease around the world. Paediatr Respir Rev. 2014 Mar;15(1):4-12. doi: 10.1016/j.prrv.2013.11.003. Epub 2013 Nov 15. PMID 24361300
- [Background] Steinberg MH, Chui DH, Dover GJ, Sebastiani P, Alsultan A. Fetal hemoglobin in sickle cell anemia: a glass half full? Blood. 2014 Jan 23;123(4):481-5. doi: 10.1182/blood-2013-09-528067. Epub 2013 Nov 12. PMID 24222332